CLINICAL TRIAL: NCT01265563
Title: Correction of Glutathione Deficiency for Treatment of Diabetic Nephropathy
Brief Title: N-Acetylcysteine and Milk Thistle for Treatment of Diabetic Nephropathy
Acronym: CGDN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CLIN-004-10S; 1R21AT004490-01A1 (NIH); VA 1I01CX000264-01A2 (Registry Identifier: VA)
Record Dates: First submitted 2010-12-10; First posted 2010-12-23 (Estimated); Results first posted 2017-03-31 (Actual); Last update posted 2018-10-19 (Actual); Status verified 2018-09

CONDITIONS: Diabetic Nephropathy; Proteinuria; Oxidative Stress
Keywords: silymarin; glutathione; diabetic nephropathies; oxidative stress; N-acetylcysteine; protein tholation
MeSH Terms: conditions — Diabetic Nephropathies; Proteinuria

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- NAC placebo and Silibin placebo (Placebo Comparator): Drug: N-acetylcysteine placebo and Drug: Silibin placebo
  Interventions: Drug: N-acetylcysteine placebo and silibin placebo
- NAC active and Silibin placebo (Experimental): Drug: N-acetylcysteine and Drug: Silibin placebo
  Interventions: Drug: N-acetylcysteine active and silibin placebo
- NAC placebo and Silibin active (Experimental): Drug: N-acetylcysteine placebo and Drug: Silibin active
  Interventions: Drug: N-acetylcysteine placebo and silibin active
- NAC active and Silibin active (Experimental): Drug: N-acetylcysteine active and Drug: Silibin active
  Interventions: Drug: N-acetylcysteine active and silibin active
- NAC active and High-dose Silibin active (Experimental): Drug: N-acetylcysteine active and Drug: Silibin higher dose active
  Interventions: Drug: N-acetylcysteine active + high-dose silibin active

INTERVENTIONS:
Drug: N-acetylcysteine placebo and silibin placebo — Dietary Supplement: N-acetylcysteine placebo excipient and silibin placebo orally twice daily for three months
  Other Names: NAC placebo, Silibin-phosphatidylcholine placebo, Siliphos placebo
  Arms: NAC placebo and Silibin placebo
Drug: N-acetylcysteine active and silibin placebo — Dietary Supplement: N-acetylcysteine 600 mg orally twice daily and silibin placebo orally twice a day for three months
  Other Names: NAC, Silibin-phosphatidylcholine placebo, Siliphos placebo
  Arms: NAC active and Silibin placebo
Drug: N-acetylcysteine placebo and silibin active — Dietary Supplement: silibin 480 mg orally twice daily and N-acetylcysteine placebo orally twice a day for three months
  Other Names: NAC Placebo, Silibin-phosphatidylcholine, Siliphos
  Arms: NAC placebo and Silibin active
Drug: N-acetylcysteine active and silibin active — Dietary Supplement: N-acetylcysteine 600 mg orally twice daily and silibin 480 mg orally twice daily for three months
  Other Names: NAC, Silibin-phosphatidylcholine, Siliphos
  Arms: NAC active and Silibin active
Drug: N-acetylcysteine active + high-dose silibin active — Dietary Supplement: N-acetylcysteine 600 mg orally twice daily and silibin 960 mg orally twice daily for three months
  Other Names: NAC, Silibin-phosphatidylcholine, Siliphos
  Arms: NAC active and High-dose Silibin active

SUMMARY:
The study is done to find out whether the combined use of the nutritional supplements N-acetylcysteine and Siliphos (milk thistle extract) corrects the shedding of urine protein and oxidative damage (damage to cells and organs often compared to fast aging) in patients with Type 2 Diabetes Mellitus (T2DM) and diabetic kidney disease.

DETAILED DESCRIPTION:
Oxidative stress and glutathione (GSH) imbalance are major contributors to the pathogenesis of diabetic nephropathy. Current options for the treatment of oxidative stress in diabetic nephropathy are limited and only partially effective, thus interest in the development of new strategies is high.

The study intends to test the hypothesis that combined oral supplementation of the antioxidants N-acetylcysteine (NAC) and milk thistle flavonolignan silibin (as silibin-phosphatidylcholine) will reduce proteinuria and urinary and systemic manifestations of oxidative stress and inflammation, which are characteristically observed in patients with T2DM and related nephropathy. The investigators expect these effects to be achieved with minimal or no side effects, and with good patient tolerance.

The trial is designed as a two-center, double-blind, placebo-controlled, randomized, modified-factorial dose-ranging design, five-arm pilot study in patients with Type 2 diabetes mellitus and advanced diabetic nephropathy with proteinuria.

Intervention consists of three-month oral administration of NAC, silibin, and/or respective placebos for three months. Subjects are randomized to the following five intervention arms: (A) placebo; (B) NAC; (C) silibin; (D) NAC + silibin; and (E) NAC + double-dose silibin.

The primary outcome measure is urinary excretion of albumin, a marker of glomerular injury. Secondary outcome measures are alpha-1 microglobulin, a marker of tubular injury, and urinary excretion of inflammatory cytokines and C-C chemokines, i.e. markers of renal inflammation. In addition, peripheral blood monocytes from the same patients are analyzed for GSH content and activity of GSH metabolizing enzymes. All outcome measures are monitored in relation to both treatment allocation and prevalent blood and urine levels of the active treatment. Safety and tolerability of this combination treatment are monitored throughout the trial.

ELIGIBILITY:
Inclusion Criteria:

* Males or females age 18-76 years old
* Type 2 diabetes mellitus
* Diabetic nephropathy, as defined by:

  * estimated GFR between 60 and 15 ml/min
  * presence of proteinuria
* Current medical treatment with low dose aspirin
* Treatment of hypertension with (but not limited to):

  * one diuretic
  * one beta-blocker
  * and one medication from the classes Angiotensin Receptor Blockers (ARBs) or Angiotensin Converting Enzyme inhibitors (ACE-I)
* Treatment of hyperglycemia with (but not limited to) glipizide and the medication class insulin
* Treatment of hypercholesterolemia with (but not limited to) one medication from the class statins

Exclusion Criteria:

* Type 1 diabetes mellitus
* Glycosylated hemoglobin (HbA1C) > 10%
* >20% variation in estimated GFR, during last 6 months
* Systolic Blood Pressure >170 mmHg or Diastolic Blood Pressure >100 mmHg on medications
* Other secondary forms of hypertension (endocrine, renovascular)
* History of intolerance to:

  * Both ACE-I and ARBs
  * The investigational supplements
  * Iodinated radiologic contrast material
* Known non diabetic renal disease
* or history of solid organ transplantation
* Hepatitis virus or Human Immunodeficiency virus infections
* Use of one of the following medications within 2 months prior to enrollment in the study:

  * Metformin
  * Thiazolidinediones (pioglitazone or rosiglitazone)
  * Phenytoin
  * Warfarin
  * Prescription-grade vitamin E, vitamin C, systemic steroids, and/or non-steroidal anti-inflammatory agents
  * Over-the-counter vitamin E, vitamin C, and/or non-steroidal anti-inflammatory agents
  * Over-the-counter antioxidants supplements including:

    * Lipoic acid
    * Coenzyme Q10
    * N-acetyl-cysteine (NAC)
    * Glutathione (GSH)
    * Chromium
    * Fish-oil extracts (omega-3 fatty acids)
    * Soy extracts (isoflavones)
    * Milk thistle extract (silymarin)
    * Green-tea preparations
    * Pomegranate extracts
    * Grape extracts
    * Prickly pear extract
* Active coronary artery disease or cerebral vascular disease within 3 months prior to signing the informed consent
* Hepatic dysfunction as defined by abnormal total bilirubin or liver enzymes (ALT, AST) >2 times upper limit of normal range
* Active malignancy
* History of drug or alcohol dependency
* Psychiatric or neurological condition, preventing aware consent to the study and/or adherence to the study protocol
* Unwillingness to practice birth control throughout the study
* Participation to another clinical study within 1 month prior to signing the informed consent form
* Planned move to outside the study area, surgery or radiographic studies utilizing iodine-based contrast material within the next one year

Ages: 18 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2011-01; Primary Completion 2015-02 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Fanti, MD, Principal Investigator — South Texas Health Care System, San Antonio, TX
Locations (1):
- South Texas Health Care System, San Antonio, TX, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Debnath S, Thameem F, Alves T, Nolen J, Al-Shahrouri H, Bansal S, Abboud HE, Fanti P. Diabetic nephropathy among Mexican Americans. Clin Nephrol. 2012 Apr;77(4):332-44. doi: 10.5414/cn107487. PMID 22445478
- [Background] Giustarini D, Dalle-Donne I, Milzani A, Fanti P, Rossi R. Analysis of GSH and GSSG after derivatization with N-ethylmaleimide. Nat Protoc. 2013 Sep;8(9):1660-9. doi: 10.1038/nprot.2013.095. Epub 2013 Aug 1. PMID 23928499
- [Result] Khazim K, Giustarini D, Rossi R, Verkaik D, Cornell JE, Cunningham SE, Mohammad M, Trochta K, Lorenzo C, Folli F, Bansal S, Fanti P. Glutathione redox potential is low and glutathionylated and cysteinylated hemoglobin levels are elevated in maintenance hemodialysis patients. Transl Res. 2013 Jul;162(1):16-25. doi: 10.1016/j.trsl.2012.12.014. Epub 2013 Jan 17. PMID 23333585
- [Result] Cunningham SE, Verkaik D, Gross G, Khazim K, Hirachan P, Agarwal G, Lorenzo C, Matteucci E, Bansal S, Fanti P. Comparison of Nutrition Profile and Diet Record Between Veteran and Nonveteran End-Stage Renal Disease Patients Receiving Hemodialysis in Veterans Affairs and Community Clinics in Metropolitan South-Central Texas. Nutr Clin Pract. 2015 Oct;30(5):698-708. doi: 10.1177/0884533615575046. Epub 2015 Apr 21. PMID 25899538
- [Result] Fanti P, Giustarini D, Rossi R, Cunningham SE, Folli F, Khazim K, Cornell J, Matteucci E, Bansal S. Dietary Intake of Proteins and Calories Is Inversely Associated With The Oxidation State of Plasma Thiols in End-Stage Renal Disease Patients. J Ren Nutr. 2015 Nov;25(6):494-503. doi: 10.1053/j.jrn.2015.06.003. Epub 2015 Jul 31. PMID 26235932
- [Result] Giustarini D, Galvagni F, Orlandini M, Fanti P, Rossi R. Immediate stabilization of human blood for delayed quantification of endogenous thiols and disulfides. J Chromatogr B Analyt Technol Biomed Life Sci. 2016 Apr 15;1019:51-8. doi: 10.1016/j.jchromb.2016.02.009. Epub 2016 Feb 8. PMID 26896310
- [Result] Khazim K, Gorin Y, Cavaglieri RC, Abboud HE, Fanti P. The antioxidant silybin prevents high glucose-induced oxidative stress and podocyte injury in vitro and in vivo. Am J Physiol Renal Physiol. 2013 Sep 1;305(5):F691-700. doi: 10.1152/ajprenal.00028.2013. Epub 2013 Jun 26. PMID 23804455

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 213 subjects met the inclusion criteria on screening from 2 clinic locations: VA and University Hospital Renal clinics.Many had exclusion criteria and few refused to participate. 108 subjects finally enrolled in the study.
Pre-assignment Details: During Run-in phase before randomization to the experimental arms, 4 subjects were excluded due to hospitalization for various reasons and 26 were excluded due to issues with transportation or sickness in the family or themselves.
Groups:
- NAC Placebo + Silibin Placebo: N-acetylcysteine placebo + silibin placebo Dietary Supplement: N-acetylcysteine placebo excipient orally twice daily for three months Other Name: NAC placebo Dietary Supplement: silibin placebo excipient orally twice daily for three months Other Name: silibin-phosphatidylcholine placebo, Siliphos placebo
  N-acetylcysteine placebo + silibin placebo: Dietary Supplement: N-acetylcysteine placebo excipient orally twice daily for three months
- NAC Active + Silibin Placebo: N-acetylcysteine active + silibin placebo Dietary Supplement: N-acetylcysteine 600 mg orally twice daily for three months Other Name: NAC Dietary Supplement: silibin placebo excipient orally twice daily for three months Other Name: silibin-phosphatidylcholine placebo, Siliphos placebo
  N-acetylcysteine active + silibin placebo: Dietary Supplement: N-acetylcysteine 600 mg orally twice daily for three months
- NAC Placebo + Silibin Active: N-acetylcysteine placebo + silibin active Dietary Supplement: silibin 480 mg orally twice daily for three months Other Name: silibin-phosphatidylcholine, Siliphos Dietary Supplement: N-acetylcysteine placebo excipient orally twice daily for three months Other Name: NAC placebo Dietary Supplement: silibin placebo excipient orally twice daily for three months Other Name: silibin-phosphatidylcholine placebo, Siliphos placebo
  N-acetylcysteine placebo + silibin active: Dietary Supplement: silibin 480 mg orally twice daily for three months
  * (Other Name) Silibin-phosphatidylcholine placebo, Siliphos placebo
  * (Other Name) NAC placebo Dietary Supplement: silibin placebo excipient orally twice daily for three months
- NAC Active + Silibin Active: N-acetylcysteine active + silibin active Dietary Supplement: N-acetylcysteine 600 mg orally twice daily for three months Other Name: NAC Dietary Supplement: silibin 480 mg orally twice daily for three months Other Name: silibin-phosphatidylcholine, Siliphos Dietary Supplement: silibin placebo excipient orally twice daily for three months Other Name: silibin-phosphatidylcholine placebo, Siliphos placebo
  N-acetylcysteine active + silibin active: Dietary Supplement: N-acetylcysteine 600 mg orally twice daily for three months
  * (Other Name): NAC Dietary Supplement: silibin 480 mg orally twice daily for three months Silibin-phosphatidylcholine, Siliphos Dietary Supplement: silibin placebo excipient orally twice daily for three months
  * (Other Name): Silibin-phosphatidylcholine, Siliphos Dietary Supplement: silibin placebo excipient orally twice daily for three months
- NAC Active + High Dose Silibin Active: N-acetylcysteine active + high-dose silibin active Dietary Supplement: N-acetylcysteine 600 mg orally twice daily for three months Other Name: NAC Dietary Supplement: high-dose silibin 960 mg orally twice daily for three months Other Name: silibin-phosphatidylcholine, Siliphos
  N-acetylcysteine active + high-dose silibin active: Dietary Supplement: N-acetylcysteine 600 mg orally twice daily for three months
Period: Overall Study
Arm/Group | NAC Placebo + Silibin Placebo | NAC Active + Silibin Placebo | NAC Placebo + Silibin Active | NAC Active + Silibin Active | NAC Active + High Dose Silibin Active
Started | 16 | 13 | 17 | 16 | 16
Completed | 16 | 12 | 16 | 16 | 14
Not Completed | 0 | 1 | 1 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- NAC Placebo and Silibin Placebo: N-acetylcysteine placebo + silibin placebo Dietary Supplement: N-acetylcysteine placebo excipient orally twice daily for three months Other Name: NAC placebo Dietary Supplement: silibin placebo excipient orally twice daily for three months Other Name: silibin-phosphatidylcholine placebo, Siliphos placebo
  N-acetylcysteine placebo + silibin placebo: Dietary Supplement: N-acetylcysteine placebo excipient orally twice daily for three months
- NAC Active and Silibin Placebo: N-acetylcysteine active + silibin placebo Dietary Supplement: N-acetylcysteine 600 mg orally twice daily for three months Other Name: NAC Dietary Supplement: silibin placebo excipient orally twice daily for three months Other Name: silibin-phosphatidylcholine placebo, Siliphos placebo
  N-acetylcysteine active + silibin placebo: Dietary Supplement: N-acetylcysteine 600 mg orally twice daily for three months
- NAC Placebo and Silibin Active: N-acetylcysteine placebo + silibin active Dietary Supplement: silibin 480 mg orally twice daily for three months Other Name: silibin-phosphatidylcholine, Siliphos Dietary Supplement: N-acetylcysteine placebo excipient orally twice daily for three months Other Name: NAC placebo Dietary Supplement: silibin placebo excipient orally twice daily for three months Other Name: silibin-phosphatidylcholine placebo, Siliphos placebo
  N-acetylcysteine placebo + silibin active: Dietary Supplement: silibin 480 mg orally twice daily for three months
  * (Other Name) Silibin-phosphatidylcholine placebo, Siliphos placebo
  * (Other Name) NAC placebo Dietary Supplement: silibin placebo excipient orally twice daily for three months
- NAC Active and Silibin Active: N-acetylcysteine active + silibin active Dietary Supplement: N-acetylcysteine 600 mg orally twice daily for three months Other Name: NAC Dietary Supplement: silibin 480 mg orally twice daily for three months Other Name: silibin-phosphatidylcholine, Siliphos Dietary Supplement: silibin placebo excipient orally twice daily for three months Other Name: silibin-phosphatidylcholine placebo, Siliphos placebo
  N-acetylcysteine active + silibin active: Dietary Supplement: N-acetylcysteine 600 mg orally twice daily for three months
  * (Other Name): NAC Dietary Supplement: silibin 480 mg orally twice daily for three months Silibin-phosphatidylcholine, Siliphos Dietary Supplement: silibin placebo excipient orally twice daily for three months
  * (Other Name): Silibin-phosphatidylcholine, Siliphos Dietary Supplement: silibin placebo excipient orally twice daily for three months
- NAC Active and High-dose Silibin Active: N-acetylcysteine active + high-dose silibin active Dietary Supplement: N-acetylcysteine 600 mg orally twice daily for three months Other Name: NAC Dietary Supplement: high-dose silibin 960 mg orally twice daily for three months Other Name: silibin-phosphatidylcholine, Siliphos
  N-acetylcysteine active + high-dose silibin active: Dietary Supplement: N-acetylcysteine 600 mg orally twice daily for three months
- Total: Total of all reporting groups
Arm/Group | NAC Placebo and Silibin Placebo | NAC Active and Silibin Placebo | NAC Placebo and Silibin Active | NAC Active and Silibin Active | NAC Active and High-dose Silibin Active | Total
Number analyzed (Participants) | 16 | 13 | 17 | 16 | 16 | 78
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 65.3 (5.74) | 64 (6.4) | 61.9 (8.39) | 64.81 (8.113) | 59.56 (7.78) | 63.09 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 0 | 2 | 2 | 7
  Male | 15 | 11 | 17 | 14 | 14 | 71
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 0 | 1
  Black or African American | 1 | 1 | 1 | 1 | 1 | 5
  White | 15 | 12 | 15 | 14 | 15 | 71
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 1
BMI [Mean (Standard Deviation); unit: kg/M^2] | 30.21 (9.28) | 39.9 (9.17) | 35.86 (8.63) | 35.65 (5.16) | 35.72 (7.5) | 35.31 (7.67)
Systolic BP [Mean (Standard Deviation); unit: mmHg] | 138.5 (21.76) | 125.54 (22.77) | 147.41 (16.8) | 137.13 (17.10) | 142.8 (12) | 139.15 (19.02)
Diastolic BP [Mean (Standard Deviation); unit: mmHg] | 70.44 (15.83) | 62.71 (12.63) | 77.47 (9.53) | 70.88 (8.37) | 74.25 (9.61) | 71.93 (12.08)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Urinary Albumin Excretion
Description: Urine albumin to creatinine ratio was assessed at the end of run in period and after 3 months administration of study intervention.
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: mg/g
Groups:
- NAC Active + High-dose Silibin Active: N-acetylcysteine active + high-dose silibin active Dietary Supplement: N-acetylcysteine 600 mg orally twice daily for three months Other Name: NAC Dietary Supplement: high-dose silibin 960 mg orally twice daily for three months Other Name: silibin-phosphatidylcholine, Siliphos
  N-acetylcysteine active + high-dose silibin active: Dietary Supplement: N-acetylcysteine 600 mg orally twice daily for three months
Arm/Group | NAC Placebo + Silibin Placebo | NAC Active + Silibin Placebo | NAC Placebo + Silibin Active | NAC Active + Silibin Active | NAC Active + High-dose Silibin Active
Number analyzed (Participants) | 16 | 12 | 16 | 16 | 14
mg/g | 50.5 (291.2) | -28.13 (578.32) | -4.5 (541) | 96.6 (422.4) | 353.71 (732.67)

2. Secondary Outcome: Change From Baseline in Hemoglobin-A1c
Description: Hemoglobin A1C was assessed at the end of the run in period and after 3 months of administration of study interventions. Here is delta HgA1C is reported between the two periods
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | NAC Placebo + Silibin Placebo | NAC Active + Silibin Placebo | NAC Placebo + Silibin Active | NAC Active + Silibin Active | NAC Active + High-dose Silibin Active
Number analyzed (Participants) | 16 | 12 | 16 | 16 | 14
percentage | 0.35 (0.58) | -0.18 (0.68) | 0.72 (2.91) | 0.4 (2.19) | 0.2 (1.14)

3. Secondary Outcome: Urinary Alpha-1 Microglobulin, Inflammatory Cytokines and C-C Chemokines
Description: Urinary alpha-1 microglobulin, inflammatory cytokines and C-C chemokines were never measured and analyzed.
Time Frame: Baseline and 3 months
Population: The secondary outcome measures: Urinary alpha-1 microglobulin, inflammatory cytokines and C-C chemokines could not be measured due to lack of research personnel support and change in the PI who didn't have sufficient expertise to assess these measures.
Arm/Group | NAC Placebo and Silibin Placebo | NAC Active and Silibin Placebo | NAC Placebo and Silibin Active | NAC Active and Silibin Active | NAC Active and High-dose Silibin Active
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | NAC Placebo + Silibin Placebo | NAC Active + Silibin Placebo | NAC Placebo + Silibin Active | NAC Active + Silibin Active | NAC Active + High-dose Silibin Active
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/12 | 0/16 | 0/16 | 0/14
Serious Adverse Events (participants affected / at risk) | 1/16 | 1/12 | 1/16 | 1/16 | 1/14
Other Adverse Events (participants affected / at risk) | 7/16 | 7/12 | 6/16 | 8/16 | 9/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NAC Placebo + Silibin Placebo (N=16) | NAC Active + Silibin Placebo (N=12) | NAC Placebo + Silibin Active (N=16) | NAC Active + Silibin Active (N=16) | NAC Active + High-dose Silibin Active (N=14)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 (1) | 0 | 0
Chest Pain (Cardiac disorders) | 0 | 1 (1) | 0 | 0 | 0
Motor Vehicle Accident (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 | 0 | 0 | 0
Osteomyelitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 (1) | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NAC Placebo + Silibin Placebo (N=16) | NAC Active + Silibin Placebo (N=12) | NAC Placebo + Silibin Active (N=16) | NAC Active + Silibin Active (N=16) | NAC Active + High-dose Silibin Active (N=14)
Heart burn, nausea, diarrhea, abd pain, anorexia (Gastrointestinal disorders) | 2 | 4 (4) | 2 (2) | 5 (5) | 4 (6)
Congestion, Sore throat, Myalgias (General disorders) | 1 | 0 | 3 (3) | 1 (1) | 1 (1)
Infection - soft tissue, UTI (General disorders) | 2 | 0 | 0 | 0 | 1 (1)
Vertigo (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Hypoglycemia (Endocrine disorders) | 1 | 0 | 0 | 0 | 1 (1)
AKI, hyperkalemia, Edema (Renal and urinary disorders) | 0 | 2 (3) | 0 | 1 (1) | 2 (2)
Flushing (Immune system disorders) | 0 | 1 (1) | 0 | 0 | 0
Fracture, sprain, stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 (2) | 0
Hypotension (Cardiac disorders) | 0 | 0 | 1 (1) | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No